CLINICAL TRIAL: NCT05652426
Title: The Effect of Hypoxic and Normoxic Cerebral Oximetry Levels and Oxidative Stress on Cognitive Functions After Carotid Endarterectomy
Brief Title: The Effect of Hypoxic and Normoxic Cerebral Oximetry Levels on Cognitive Functions After Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: ISuidiye
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Hypoxia; Carotid Stenosis; Cognitive Dysfunction
MeSH Terms: conditions — Hypoxia, Brain; Carotid Stenosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Basal cerebral oximetry levels between 41-60%
- Group 2: Basal cerebral oximetry levels > 61%

SUMMARY:
In this study, we investigated the effect of the capacity to cope with oxidative stress (oxidative stress response during and after clamping) in individuals with cerebral oximetry level between 40- 60 % and above 60 % and their effect on cognitive functions.

Methods: In this retrospective study, patients who were scheduled for carotid endarterectomy, examined the MOCA tests before and after the operation and collected blood samples intraoperatively were included between January 2020-2021. The time periods specified below, blood samples were taken and serums were frozen at -80 celcius all this patients. Montreal cognitive function assessment test was applied before the operation, 24 hours and 7 days after the operation. Ten mililiters venous blood samples were collected to examine the status of basal neuron specific enolase, S100B, oxydative stress parameters (HAF-1 and DAF-1) at time intervals. Time intervals as follow:

T1: Peripheral baseline measurements (blood will be taken from arterial blood sampling) + Cerebral Oxymeter levels + Montreal cognitive performance test + Modified Rankin Scale (mRS) T2: 1 minute before clamping (from peripheral and jugular vena blood sampling) + Cerebral Oxymeter levels T3: Before opening clamp(from peripheral and jugular vena blood sampling) + Cerebral Oxymeter levels T4: 24 hours after the procedure. (peripheral blood sampling) + Montreal cognitive performance test T5: 7 days after the operation. (peripheral blood sampling) + Montreal cognitive performance test + CO levels+ Modified Rankin Scale (mRS) Results: We found significantly positive corelation between cerebral oxymeter levels, oxydative stress parameters and cognitive performance tests in this six patient.

DETAILED DESCRIPTION:
In this retrospective study, patients who were scheduled for carotid endarterectomy, examined the MOCA (Montreal cognitive assesment )tests before and after the operation and collected blood samples intraoperatively were included between January 2020-2021. The time periods specified below, blood samples were taken and serums were frozen at -80 celcius all this patients. Montreal cognitive function assessment test was applied before the operation, 24 hours and 7 days after the operation. Ten mililiters venous blood samples were collected to examine the status of basal neuron specific enolase, S100B, oxydative stress parameters (HAF-1 and DAF-1) at time intervals. Time intervals as follow:

T1: Peripheral baseline measurements (blood will be taken from arterial blood sampling) + Cerebral Oxymeter levels + MoCA + Modified Rankin Scale (mRS) T2: 1 minute before clamping (from peripheral and jugular vena blood sampling) + Cerebral Oxymeter levels T3: Before opening clamp(from peripheral and jugular vena blood sampling) + Cerebral Oxymeter levels T4: 24 hours after the procedure. (peripheral blood sampling) + MoCA test T5: 7 days after the operation. (peripheral blood sampling) + MoCA + CO levels+ Modified Rankin Scale The degree of stenosis was determined according to the North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria. Written informed consent form was obtained from the patients 1 day before the operation. Basal invasive arterial blood pressure, pulse oximetry, heart rate, cerebral perfusion pressure, cerebral oximetry levels records of all patients were taken as baseline values before the operation. During the operation, serum samples were taken and 5 ml blood samples were taken from the artery (peripheral) and 5 ml from the vena jugularis interna during the operation. Blood samples were immediately centrifuged at 15000 rpm for 15 minutes and the supernatant was collected. The supernatant was immediately stored at -80 °C for further analysis of oxidative stress and other parameters. The parameters studied are: Human NSE(Neuron Specific Enolase) ELISA Kit, Neuron Specific Enolase ELISA Kit, Human S100B (S100 Calcium Binding Protein B) ELISA Kit, HIF-1α (Hypoxia Inducible Factor 1 Alpha) ELISA Kit, Human DAF(Decay Accelerating Factor) ELISA Kit.

A. General anesthesia procedure: Anesthesia induction was performed with 1-2 mg/kg propofol, 1 mcg/kg fentanyl, 0.5 mg/kg rocuronium. Anesthesia was maintained with remifentanil infusion (0.05-0.1 mcg/kg/min), 1-2% sevoflurane (1 MAC), and rocuronium. Mechanical ventilation parameters were adjusted to be within the limits of end-tidal carbon dioxide normocarby (35-45mm Hg) (mean 40 mmHg). To prevent the development of bradycardia, 1% lidocaine was applied to the internal, external and common carotid arteries by the surgical team. Following systemic intravenous (5000 IU) heparin administration, carotid arterial cross-clamp was placed with appropriate active clotting time (>200) B. Superficial and deep cervical blockade: It was done with 0.5% isobaric bupivacaine 15 ml + 2% prilocaine 5 ml.

ΔrSO2 (%) = 100 x (rSO2preclamping - rSO2baseline) / rSO2baseline Baseline rSO2 value, rSO2 measurement for each specific time point and %rSO2 change between them were continuously monitored by oximetry (Invos System 4100, Somonetics Corporation, Troy, MI, USA). The entire CEA surgical procedure was performed with the standardized technique in these 6 patients.

In the analysis phase, the patients were evaluated in 2 groups. Group 1: Basal cerebral oximetry levels between 41-60% Group 2: Basal cerebral oximetry levels > 61%

ELIGIBILITY:
Inclusion Criteria:

Patients who were scheduled for carotid endarterectomy, examined the MOCA (Montreal cognitive assesment )tests before and after the operation and collected blood samples intraoperatively were included between January 2020-2021.

Exclusion Criteria:

* Irregular diabetes mellitus
* Pregnancy
* Acute or chronic renal failure
* Liver failure
* History of previous carotid or brain trauma
* Vasculitis
* Thyroid diseases
* Adrenal insufficiency
* Patients who cannot perform cognitive function tests
* Anemia (below 10 g/dl)
* History of previous stroke in the last 6 months
* Patients with plegia in the dominant upper extremity
* Patients who will be shunted during the operation.
* Patients with vertebrobacillary arterial system or ring of Willis anomaly
* Presence of acute myocardial infarction.
* Traumatic brain injuries less than 6 months before the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled for carotid endarterectomy, examined the MOCA (Montreal cognitive assesment )tests before and after the operation and collected blood samples intraoperatively .
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Serebral biomarkers | 7 day
  To investigate the correlation of brain oxygenation with cerebral biomarkers in patients with two different basal rSO2 levels (41-60% rSO2 and above 60% rSO2) in carotid endarterectomy operations.

SECONDARY OUTCOMES:
Oxydative stress parameters | 7 day
  To investigate the correlation of brain oxygenation with oxydative stress biomarkers in patients with two different basal rSO2 levels (41-60% rSO2 and above 60% rSO2) in carotid endarterectomy operations.
Cognitive function | 7 day
  To investigate the effect of basal brain oxygenation status on postoperative cognitive function and correlation with cerebral biomarkers, oxydative stress parameters in patients with two different basal rSO2 levels (41-60% rSO2 and above 60% rSO2) in carotid endarterectomy operations.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur S Yorulmaz, Principal Investigator — Duzce University
Locations (1):
- İlknur Suidiye Yorulmaz, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heyer EJ, Sharma R, Rampersad A, Winfree CJ, Mack WJ, Solomon RA, Todd GJ, McCormick PC, McMurtry JG, Quest DO, Stern Y, Lazar RM, Connolly ES. A controlled prospective study of neuropsychological dysfunction following carotid endarterectomy. Arch Neurol. 2002 Feb;59(2):217-22. doi: 10.1001/archneur.59.2.217. PMID 11843692
- [Background] Zhang HP, Ma XD, Chen LF, Yang Y, Xu BN, Zhou DB. Cognitive Function After Carotid Endarterectomy: Early Decline and Later Recovery. Turk Neurosurg. 2016;26(6):833-839. doi: 10.5137/1019-5149.JTN.13382-14.1. PMID 27438617
- [Background] Kuzhuget R, Starodubtsev V, Ignatenko P, Starodubtseva A, Voroshilina O, Ruzankin P, Karpenko A. The role of stump pressure and cerebral oximetry in predicting ischaemic brain damage during carotid endarterectomy. Brain Inj. 2017;31(13-14):1944-1950. doi: 10.1080/02699052.2017.1347279. Epub 2017 Sep 5. PMID 28872355
- [Background] Koh MY, Powis G. Passing the baton: the HIF switch. Trends Biochem Sci. 2012 Sep;37(9):364-72. doi: 10.1016/j.tibs.2012.06.004. Epub 2012 Jul 18. PMID 22818162
- [Background] Schmid T, Zhou J, Brune B. HIF-1 and p53: communication of transcription factors under hypoxia. J Cell Mol Med. 2004 Oct-Dec;8(4):423-31. doi: 10.1111/j.1582-4934.2004.tb00467.x. PMID 15601571
- [Background] Lee JW, Bae SH, Jeong JW, Kim SH, Kim KW. Hypoxia-inducible factor (HIF-1)alpha: its protein stability and biological functions. Exp Mol Med. 2004 Feb 29;36(1):1-12. doi: 10.1038/emm.2004.1. PMID 15031665
- [Background] Hashimoto T, Shibasaki F. Hypoxia-inducible factor as an angiogenic master switch. Front Pediatr. 2015 Apr 24;3:33. doi: 10.3389/fped.2015.00033. eCollection 2015. PMID 25964891